CLINICAL TRIAL: NCT00678405
Title: Phase III Randomized Controlled Trial of a Breathlessness Intervention Service for Intractable Breathlessness.
Brief Title: Trial of a Breathlessness Intervention Service for Intractable Breathlessness
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); King's College London (Other)
Responsible Party: Dr Sara Booth, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PB-PG-0107-11134; ISRCTN04119516
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Dyspnea
Keywords: Breathlessness; Dyspnoea; Dyspnea; Palliative care; RCT; Randomised controlled trial; Lung cancer; COPD; Heart failure; Chronic respiratory disease
MeSH Terms: conditions — Dyspnea; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WLm / WLnm (Active Comparator): Best supportive care
  Interventions: Behavioral: Best supportive care (Standard Care)
- FTm / FTnm (Experimental): Breathlessness Intervention Service
  Interventions: Behavioral: Breathlessness Intervention Service

INTERVENTIONS:
Behavioral: Breathlessness Intervention Service — Breathlessness Intervention Service (BIS) consists of a clinical specialist physiotherapist & palliative care consultant. It aims to manage the symptom of breathlessness in patients with any disease (cancer & non-cancer) using a rehabilitative approach. Interventions include: evidence-based non-pharmacological interventions (psychological, social & physical); palliative care input (e.g. end of life issues, psychosocial issues, family concerns); & pharmacological review. Thus BIS seeks to enhance the self-management of breathlessness. Uniquely, care is located in clinic or in patients' own homes, as appropriate. Referrals come from medical specialists, GPs & allied health professionals (with medical consent).
  Other Names: BIS
  Arms: FTm / FTnm
Behavioral: Best supportive care (Standard Care) — Standard care: specialist outpatient appointments in secondary care (e.g. respiratory, cardiology, neurology or oncology) which may include specialist nurse input, and primary care services.
  Other Names: Standard care
  Arms: WLm / WLnm

SUMMARY:
The aim of this study is to evaluate the impact of a Breathlessness Intervention Service (BIS) on the quality of life of patients and families affected by intractable breathlessness. The questions to be addressed by this research are:

1. Is BIS more effective than standard care for patients with intractable breathlessness from advanced malignant or non-malignant disease?
2. Does it reduce patient and carer distress due to breathlessness, and increase patients' sense of mastery of the symptom?
3. What are the experiences and views of those who use BIS, their informal carers and the clinicians who refer to it?
4. Does BIS offer value for money for the NHS?

DETAILED DESCRIPTION:
Research questions:

1. Is BIS more effective than standard care for patients with intractable breathlessness from advanced malignant or non-malignant disease?
2. Does it reduce patient & carer distress due to breathlessness, & increase patients' sense of mastery of the symptom?
3. What are the experiences & views of those who use BIS, their informal carers & the clinicians who refer to it?
4. Is BIS cost-effective?

To assess changes in patient outcomes attributable to BIS, a pragmatic RCT design will be conducted using a fast-track design (design proved highly acceptable at Phase II). Analysis will focus on comparing patients who have used BIS to those who have not (yet) used BIS (the use of BIS by the control group will occur subsequent to these measurement points).

The researcher will be blinded to the allocation of respondents up until discharge/referral on from BIS for FT patients or at the end of the waiting period for CC patients. This will be achieved by the researcher conducting study recruitment & collecting baseline measures before instructing a third party (local clinical trials' nurse) to conduct randomisation & reporting of allocation (to the patient & BIS) using a random sequence of opaque envelopes previously generated by a statistician independent of BIS. Subsequently, all data will be handled using study identity numbers; group allocation identifiers will only be added at analysis. This model was used successfully in the Phase II pilot trial.

Data collected from the control group once they are in receipt of BIS (after their period on the waiting list when their group allocation was blinded to the researcher) will be treated as before/after data & not RCT data. This will allow the collection of qualitative data from this group at the midpoint of using BIS.

The two broad disease courses, malignant (m) & non-malignant (nm), will be considered separately due to their different trajectories & needs, & resultant different service models. The intervention model for patients with non-malignant disease consists of two-three visits & three telephone contacts (to patient &/or primary care staff) over a four-week period with a 16 week (from first assessment) follow up, whereas the model for patients with malignant disease consists of one visit in conjunction with a primary care professional/key worker & two telephone contacts (to patient &/or primary care staff/key worker) over a two-week period, with a six week (from first assessment) follow up . Thus, the measurement points for the disease groups will differ.

Data (quantitative/qualitative) will be collected for all respondents at baseline (t1), prior to randomisation. For those with non-malignant conditions (nm), this will be repeated for the FT group (nmFT) midway through the intervention (two weeks post commencing BIS; nmFTt2 - quantitative data only) & at the equivalent time point for the CC group (i.e. two weeks from entering the waiting list; nmCCt2 - quantitative data only), then again after discharge/referral on from BIS for the fast track group (four weeks post commencing BIS; nmFTt3) & four weeks after discharge (nmFTt5). As well as being interviewed at t1 (randomisation) & t2 (midway between randomisation & BIS - quantitative data only), the CC group (nmCC) will also be interviewed just prior to commencing BIS (nmCCt3), during BIS (two weeks post commencing BIS; nmCCt4) & then again after discharge/referral on from BIS (four weeks post commencing BIS (nmCCt5). This will allow identification of whether or not respondents in the control group deteriorated significantly whilst waiting for BIS & the impact of this on final outcomes. This model was successfully piloted at Phase II.

For those with malignant conditions (m), baseline measures (t1) will be repeated for the FT group (mFT) after discharge/referral on from BIS (two weeks post commencement of BIS; mFTt3) & two weeks after discharge (mFTt5). For the CC group (mCC) baseline measures (t1) will be repeated just prior to commencing BIS (mCCt3) & then again after discharge/referral on from BIS (two weeks post commencing BIS; mCCt5). Thus, due to the shorter time frame of the malignant service model, there would be no t2 or t4 measurement points.

Sample size is based on the existing literature & on our experiences at Phase II. The estimated standard deviation of the primary outcome measure is 2.5. In order to detect a 2-point difference in mean outcome between groups (equivalent to 0.8sd effect size) with 80% power using a t-test at the 5% level of significance, it will be necessary to recruit 26 patients per arm per disease group (trial) followed up to provide an outcome, which will now be at an earlier time point to minimize attrition. By adjusting for the baseline of the primary outcome measure in the analysis using analysis of covariance we anticipate an improvement in the precision of the estimated intervention effect. We also anticipate an improvement from the use in the trial of the NRS measure rather than the more highly variable VAS version from the pilot used in this sample size calculation. Therefore we propose to recruit 120 patients, 60 per disease group to ensure adequate power, effect size and allowance for attrition.

Analysis will be on an intention to treat basis. Primary analysis will be by analysis of covariance of the NRS at the final time-point with adjustment for baseline NRS in order to improve precision of the estimated BIS versus comparison effect. Secondary analysis will more sensitively incorporate all time-points in a repeated measures linear regression to be able to detect any differences between BIS & comparison emerging/changing over time within the initial period. All analysis will be documented prior to final data collection in an analysis plan, will be addressed with two-tailed tests & be assessed at the 5% level of significance. Effects within & between arms will be summarized using means & 95% confidence intervals. If randomised effects are similar in malignant & non-malignant groups, a combined effect will be estimated allowing a narrower overall confidence interval. Analysis will be conducted using SPSS software.

The cost of BIS for each patient will be calculated from service activity data combined with staff salary costs, plus on-costs, overheads & equipment. Information on the use of other health & social services & informal care (proxy-valued as a homecare worker) will be collected with the Client Service Receipt Inventory. This will be combined with appropriate unit cost data (Curtis & Netten, 2006) to generate service costs. Cost comparisons will be made using bootstrapping methods to account for any skewness in data distribution. Cost-effectiveness will be assessed by combining cost data with that on outcomes including quality-adjusted life years (QALYS), in the form of incremental cost-effectiveness ratio & acceptability curves. Qualitative data will be analysed using a framework approach (Ritchie & Spencer, 1993) conducted using NVivo software.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

1. appropriate referral to BIS
2. aged 18 years+
3. any patient not meeting any exclusion criteria.

Carer inclusion criteria:

1. informal carers (significant others, relatives, friends or neighbors) of Phase III RCT recruits
2. aged 18 years+
3. any carer not meeting any exclusion criteria.

Exclusion Criteria:

1. unable to give informed consent
2. previously used BIS
3. demented/confused
4. learning difficulties
5. other vulnerable groups e.g. head injury, severe trauma, mental illness
6. not meeting all inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Numerical rating Scale (NRS) for distress due to breathlessness | End of intervention (4 weeks after baseline for patients with a non-malignant diagnosis; 2 weeks after baseline for patients with malignant diagnoses)

SECONDARY OUTCOMES:
Modified BORG | As for primary outcome measure
NRS Breathlessness at best/worst | as for primary outcome measure
Dyspnoea descriptors | as for primary outcome measure
CRQ | as for primary outcome measure
EQ-5D | as for primary outcome measure
HADS | as for primary outcome measure
CSRI | as for primary outcome measure
Charlson Co-morbidity score | as for primary outcome measure
Social Functioning | as for primary outcome measure
Karnofsky | as for primary outcome measure
Experience of breathlessness and expectations/views of BIS | as for primary outcome measure
Burden interview and caregiver Appr scale | as for primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Sara Booth, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Booth S, Silvester S, Todd C. Breathlessness in cancer and chronic obstructive pulmonary disease: using a qualitative approach to describe the experience of patients and carers. Palliat Support Care. 2003 Dec;1(4):337-44. doi: 10.1017/s1478951503030499. PMID 16594223
- [Background] Booth S, Farquhar M, Gysels M, Bausewein C, Higginson IJ. The impact of a breathlessness intervention service (BIS) on the lives of patients with intractable dyspnea: a qualitative phase 1 study. Palliat Support Care. 2006 Sep;4(3):287-93. doi: 10.1017/s1478951506060366. PMID 17066970
- [Background] Booth S, Wade R. Oxygen or air for palliation of breathlessness in advanced cancer. J R Soc Med. 2003 May;96(5):215-8. doi: 10.1177/014107680309600503. No abstract available. PMID 12724429
- [Background] Booth S, Adams L. The shuttle walking test: a reproducible method for evaluating the impact of shortness of breath on functional capacity in patients with advanced cancer. Thorax. 2001 Feb;56(2):146-50. doi: 10.1136/thorax.56.2.146. PMID 11209105
- [Background] Booth S. The management of dyspnoea in advanced cancer. Hosp Med. 1998 May;59(5):348-9. No abstract available. PMID 9722382
- [Background] Bausewein C, Farquhar M, Booth S, Gysels M, Higginson IJ. Measurement of breathlessness in advanced disease: a systematic review. Respir Med. 2007 Mar;101(3):399-410. doi: 10.1016/j.rmed.2006.07.003. Epub 2006 Aug 17. PMID 16914301
- [Background] Bausewein C, Booth S, Gysels M, Higginson I. Non-pharmacological interventions for breathlessness in advanced stages of malignant and non-malignant diseases. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD005623. doi: 10.1002/14651858.CD005623.pub2. PMID 18425927
- [Background] Booth S, Wade R, Johnson M, Kite S, Swannick M, Anderson H; Expert Working Group of the Scientific Committee of the Association of Palliative Medicine. The use of oxygen in the palliation of breathlessness. A report of the expert working group of the Scientific Committee of the Association of Palliative Medicine. Respir Med. 2004 Jan;98(1):66-77. doi: 10.1016/j.rmed.2003.08.008. PMID 14959816
- [Background] Bredin M, Corner J, Krishnasamy M, Plant H, Bailey C, A'Hern R. Multicentre randomised controlled trial of nursing intervention for breathlessness in patients with lung cancer. BMJ. 1999 Apr 3;318(7188):901-4. doi: 10.1136/bmj.318.7188.901. PMID 10102851
- [Background] Corner J, Plant H, A'Hern R, Bailey C. Non-pharmacological intervention for breathlessness in lung cancer. Palliat Med. 1996 Oct;10(4):299-305. doi: 10.1177/026921639601000405. PMID 8931065
- [Background] Farquhar MC, Higginson IJ, Fagan P, Booth S. The feasibility of a single-blinded fast-track pragmatic randomised controlled trial of a complex intervention for breathlessness in advanced disease. BMC Palliat Care. 2009 Jul 7;8:9. doi: 10.1186/1472-684X-8-9. PMID 19583857
- [Background] Farquhar M, Higginson IJ, Booth S. Fast-track trials in palliative care: an alternative randomized controlled trial design. J Palliat Med. 2009 Mar;12(3):213. doi: 10.1089/jpm.2008.0267. No abstract available. PMID 19254192
- [Derived] Farquhar MC, Prevost AT, McCrone P, Brafman-Price B, Bentley A, Higginson IJ, Todd CJ, Booth S. The clinical and cost effectiveness of a Breathlessness Intervention Service for patients with advanced non-malignant disease and their informal carers: mixed findings of a mixed method randomised controlled trial. Trials. 2016 Apr 4;17:185. doi: 10.1186/s13063-016-1304-6. PMID 27044249
- [Derived] Javadzadeh S, Chowienczyk S, Booth S, Farquhar M. Comparison of respiratory health-related quality of life in patients with intractable breathlessness due to advanced cancer or advanced COPD. BMJ Support Palliat Care. 2016 Mar;6(1):105-8. doi: 10.1136/bmjspcare-2015-000949. Epub 2015 Dec 18. PMID 26685116
- [Derived] Farquhar MC, Prevost AT, McCrone P, Brafman-Price B, Bentley A, Higginson IJ, Todd C, Booth S. Is a specialist breathlessness service more effective and cost-effective for patients with advanced cancer and their carers than standard care? Findings of a mixed-method randomised controlled trial. BMC Med. 2014 Oct 31;12:194. doi: 10.1186/s12916-014-0194-2. PMID 25358424
- [Derived] Farquhar MC, Prevost AT, McCrone P, Higginson IJ, Gray J, Brafman-Kennedy B, Booth S. Study protocol: Phase III single-blinded fast-track pragmatic randomised controlled trial of a complex intervention for breathlessness in advanced disease. Trials. 2011 May 20;12:130. doi: 10.1186/1745-6215-12-130. PMID 21599896